CLINICAL TRIAL: NCT03604471
Title: Lipid-lowering Therapy Individualization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Laure Elens, Professor, Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/26OCT/471
Record Dates: First submitted 2018-06-27; First posted 2018-07-27 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atorvastatin (Other): All patients using atorvastatin at any dose (usually ranging from 5 to 80 mg once-daily).
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Blood sampling for atorvastatin quantification and pharmacogenetic analysis.

SUMMARY:
This clinical study will explore individual factors influencing statin pharmacokinetics in a cohort of 150 patients treated with atorvastatin.

DETAILED DESCRIPTION:
Atorvastatin is widely prescribed for the treatment of hypercholesterolemia to prevent the risk of cardiovascular diseases, a leading death cause in industrialized countries. There exists considerable inter-individual variability in response to statins, reflected by differences in lipid-lowering effect or risk of presenting adverse drug reaction; mainly myotoxicity. A plethora of different factors (demographic, genetic, physiopathologic, environmental...) have been tested to explain this variability but it lacks of pharmacokinetic (PK) data and/or replications of observations are rare and results remain inconclusive, probably because of non-adapted designs and no-clear driven-hypothesis but also due to a lack of scientific rationale and deep mechanistic understanding. This clinical study will explore individual factors influencing statin PK in a cohort of 150 patients treated with atorvastatin. The collection of meticulous clinical PK data and a rigorous statistical analysis will allow quantifying the effect of each identified parameter on statin PK and eventually, defining a population-based PK model taking into account the combined effect of all covariates in a quantitative approach. This innovative prospectively designed clinical study will ultimately allow predicting atorvastatin PK fluctuations and anticipating any inadequate dosing in clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with atorvastatin (any dose)

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Atorvastatin population pharmacokinetics | 18 months
  Concentrations of atorvastatin acid (pmol/ml) will be measured by HPLC-MS using sparse samples obtained over the entire study period. Data will be pooled and analyzed using population pharmacokinetic modeling. The reported pharmacokinetic parameters will depend on the type of model that best fits the data.
Atorvastatin metabolites population pharmacokinetics | 18 months
  Concentrations of ortho-hydroxyatorvastatin (pmol/ml), para-hydroxyatorvastatin (pmol/ml) and atorvastatin lactone (pmol/ml) will be measured by HPLC-MS using sparse samples obtained over the entire study period. Data will be pooled and analyzed using population pharmacokinetic modeling. The reported pharmacokinetic parameters will depend on the type of model that best fits the data.

SECONDARY OUTCOMES:
Cholesterol | 18 months
  Measurement of total cholesterol, LDL cholesterol and HDL cholesterol at each visit
Creatine kinase | 18 months
  Measurement of creatine kinase at each visit
Occurrence of adverse drug events | 18 months
  Reports of adverse drug events will be recorded at each visit using a standardized questionnaire that includes the following categories : muscle cramps (grade 1 to 5), muscle pain (graded 1 to 5), rhabdomyolysis, gastro-intestinal side effects (Nauseas, diarrhea or vomitus), other side effects.
Pharmacogene genotype | 18 months
  Patients will be genotyped for single nucleotide polymorphisms of interest in the following genes : ABCB1, ABCC1, ABCC2, ABCC4, ABCC5, ABCG2, CYP3A4, CYP3A5, NR1I2, POR, PPARalpha, SLCO1B1, SLCO2B1, SLCO3A1.
Triglycerides | 18 months
  Measurement of triglyceride levels at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Balligand, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No